CLINICAL TRIAL: NCT06344156
Title: Adjuvant Therapy of Neoantigen Vaccine Plus Anti-PD1 and Chemotherapy in Patients With Resected Pancreatic Cancer
Brief Title: Neoantigen Vaccine Plus Anti-PD1 and Chemotherapy as an Adjuvant Therapy for Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHANT-231
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer; Adjuvant Therapy
Keywords: Pancreatic Cancer; Neoantigen; Adjuvant therapy; Safety; Clinical efficacy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoantigen Vaccine Plus Anti-PD1 and Chemotherapy (Experimental): (1)8 cycles of Gemcitabine +capecitabine (Gemcitabine d1,8 ,Capecitabine d1-14 q3w）；（2） two 200 mg intravenous dose of tislelizumab (d1,q3w)（3）five intravenous doses of neoantigen vaccines given as priming doses(d1,8,22,36,50）and two booster dose(d80,d110)
  Interventions: Drug: Neoantigen Vaccine Plus Anti-PD1 and Chemotherapy

INTERVENTIONS:
Drug: Neoantigen Vaccine Plus Anti-PD1 and Chemotherapy — Gemcitabine +capecitabine, tislelizumab, neoantigen vaccines

SUMMARY:
The aim of this single center, single arm and prospective study is to explore the safety and efficacy of Neoantigen Vaccine Plus Anti-PD1 and Chemotherapy in postoperative adjuvant treatment of Pancreatic Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and age ≤75 years.
2. ECOG score 0-1.
3. Patients with histologically confirmed pancreatic ductal adenocarcinoma, R0 resection, stage I-III, not receiving neoadjuvant therapy.
4. Adequate bone marrow and organ function:
5. Patients of childbearing potential must take appropriate precautions prior to enrollment and during the study.
6. Signed informed consent.
7. Ability to comply with the study protocol and follow-up.

Exclusion Criteria:

1. Received antitumor chemotherapy, radiation therapy, or immunotherapy within 2 weeks prior to first vaccination.
2. The patient has a history of other tumors, except for cervical cancer in situ, treated squamous cell carcinoma or urothelial tumors (Ta and TIS), or other malignancies that have been treated with curative intent (at least 5 years prior to enrollment).
3. Uncontrollable comorbidities, including but not limited to active bacterial or fungal infections, symptomatic congestive heart failure, unstable angina, arrhythmias.
4. HIV infection or active hepatitis B (HBV DNA≥500IU/ml), hepatitis C.
5. Uncontrolled coronary artery disease or asthma, uncontrolled cerebrovascular disease, or other conditions deemed ineligible by the investigator.
6. Uncontrollable comorbidities, including but not limited to active bacterial or fungal infections, congestive heart failure, unstable angina, arrhythmias, etc;
7. Patients with autoimmune diseases or immunodeficiencies being treated with immunosuppressive drugs.
8. Pregnant or lactating women.
9. Vaccination with other preventive vaccines within 4 weeks before the first administration or planned during the study period, including within 8 weeks after the last vaccination.
10. Those who have had a severe allergic reaction to vaccines for other infectious diseases in the past.
11. Those who may be allergic to the investigational product or any of its excipients.
12. Substance abuse or inability to undergo immunotherapy due to clinical, psychological, or social factors.
13. Significant weight loss (≥10%) within 6 weeks prior to enrollment.
14. Any uncertain factors that may affect patient safety or compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
18-month RFS | through study completion, an average of 2 year
  defined recurrence as new lesions on the basis of response evaluation criteria in solid tumours (v.1.1), and RFS from either the date of surgery (RFS) or from the date of the last neoantigen vaccine priming dose to the date of recurrence or death, whichever occurred first.
Incidence of Treatment-Related Adverse Events [Safety and Tolerability] | 3 months after the last administration of neoantigen vaccine
  Defined by treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
18-month OS | through study completion, an average of 3 year
  defined OS from the date of surgery to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: zhong Wu, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes